CLINICAL TRIAL: NCT02863783
Title: Pilot Trial of Endoscopic Ultrasound Guided Coil Placement to Facilitate Intraoperative Assessment of Pancreas Tumors
Brief Title: EUS Fiducial for Pancreas Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Associate Professor of Clinical Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00032
Record Dates: First submitted 2016-07-31; First posted 2016-08-11 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fiducial Placement (Experimental): EUS with Fiducial Placement into Tumor
  Interventions: Device: EUS with Fiducial

INTERVENTIONS:
Device: EUS with Fiducial — EUS will be used to place fiducial into pancreas tumor at time of biopsy

SUMMARY:
RATIONALE: Pancreas tumor localization makes minimally invasive surgical resection of pancreas tumors very challenging. Recently, an endoscopic ultrasound needle system has been developed which enables fiducial coils to be placed at the precise site of biopsy.

INTERVENTION: At time of EUS guided biopsy the fine needle fiducial device will be used to place fiducials in the tumor. During surgery we will assess whether it improves tumor visualization.

OBJECTIVES: We aim to determine the feasibility to use EUS guided fiducials placement to mark pancreas tumors in 20 patients and to assess whether the fiducials impact tumor visualization during pancreas surgery.

STUDY POPULATION: Patients with pancreas adenocarcinoma or neuroendocrine lesions.

STUDY ENDPOINTS: The main outcome will be to assess whether the coil may be successfully placed during EUS and whether they impact tumor visualization during surgery FOLLOW UP and ANALYSIS: Patients will be assessed at the time of EUS and surgery. This is a pilot analysis with the intention to assess feasibility and to gather data to power larger trials.

DETAILED DESCRIPTION:
Minimally invasive pancreatic surgery diminishes the morbidity and mortality of the potentially curative procedures. However precise targeting of small adenocarcinomas and neuroendocrine tumors is challenging.

Given safety, precision, and ease EUS guided pancreatic fiducial placement has emerged as a favored method to mark tumors for radiation therapy. The experimental aspect of this procedure is gauge whether EUS guided fiducial placement improves the intraoperative assessment of pancreas tumors. We will use the recently introduced (FDA approved) Beacon EUS guided fiducial system to perform placement. The fiducial will not alter the surgical plan in this study. However, the relative ability to detect the marker during standard pancreatic surgery will help to inform whether this strategy may be used in improve future approaches to pancreas surgery.

The study will be a prospective trial. All EUS will be performed as part of standard clinical care.

Conventional EUS+FNA The linear array echoendoscope will be used to identify the pancreas adenocarcinoma and neuroendocrine tumors. The Beacon EUS system/delivery sheath will be passed and fine needle aspiration performed to confirm cytology. This is required for standard clinical care. The delivery sheath will be left in place. The cytologist will perform bedside interpretation as is standard clinical care.

EUS guided coil injection If adenocarcinoma or neuroendocrine tumor is confirmed by fine needle aspiration the fine needle fiducial accessory will be passed through the delivery sheath (whose position on the tumor is now "biopsy confirmed" and 1-3 fiducials (coil type) will be introduced into the lesion. This process will be guided by EUS which is being performed for standard clinical care. Fluoroscopy not be utilized.

Pancreas Surgery: At time of surgery the experimental component is that it will be gauged whether the fiducial impacts the ability to assess the tumor relative to lesions of comparable size. Whether the fiducial improves or does not improve assessment will be scaled on a 1-10 scale where 5 is the standard ease of detection of similarly sized tumors (without fiducials) based on the attending surgeon's experience.

However, the fiducial will not be used to target the lesion or alter the surgical plan. The surgical plan will be based on preoperative clinical imaging, intraoperative findings, and intraoperative ultrasound (standard clinical care). The research coordinator will be present during surgery to facilitate timely acquisition of data. In some cases patient are deemed to not be resection candidates at the time of surgery if for example unexpected metastasis are found. The EUS guided fiducial placement will have no bearing on whether resection is done or not.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing endoscopic ultrasound for preoperative evaluation before planned pancreatic surgery for suspected adenocarcinoma and neuroendocrine tumors will be eligible. Rapid onsite evaluation is performed for all pancreas EUS as part of standard procedures. In this process the cytologist examines the cells and makes a determination whether the aspirate contains malignant or benign tissue. Fiducials will only be placed if cytologic confirmation of malignancy at the site is obtained.

Tumors of sizes 5mm-4cm will be eligible as there may be benefit in marking small tumors given difficulty finding them with intraoperative ultrasound. Moderately large pancreas tumors may also cause fibrosis which makes identification for resection difficult. Coil placement in regions of cytologically confirmed malignant cells may be helpful. Fiducial markers will only be placed if the initial evaluation (abdominal computed tomography or magnetic resonance imaging) indicates resectability. If finding of nonresectability (i.e. liver metastasis) are seen on EUS then fiducials will not be placed.

Exclusion Criteria:

* 1) Patients with INR >1.5 2) Platelet county <100 3) Metal allergy 4) Pregnant 5) <18 years of age 6) Patients with pancreatic lymphoma will also be excluded as this is treated with chemotherapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The Proportion of patients in which the fiducial was successfully placed/total patients in which fiducial attempted | 3 months
  the primary outcome will be to assess whether the coil may be successfully placed. This will be reported as the proportion of patients in which the fiducial was successfully placed/total patients in which fiducial attempted.
Relative Ease of Detection of the Tumor with Fiducial | 3 months
  A co-primary outcome will be to assess whether the coil may detected at time of surgery. The proportion of patients in whom the fiducial may be easily detected will also be reported. The relative ease of detection of the tumor (with fiducial) will be compared to the ease of detection of similar sized tumors without the fiducial. A QUESTIONNAIRE will be used in which each of detection by the attending surgeon will be recorded with 5 being each of detection of similar (histology/size) tumor without fiducial.

SECONDARY OUTCOMES:
Pancreatitis, abdominal pain, infection, bleeding following placement. | 3 months
  all complications including acute pancreatitis, abdominal pain, infection, bleeding following EUS guided fiducial placement will be recorded and reported. This will also be reported as the proportion of patients who develop a complication divided by total patients. Individual types of complications will be similarly reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Park WG, Yan BM, Schellenberg D, Kim J, Chang DT, Koong A, Patalano C, Van Dam J. EUS-guided gold fiducial insertion for image-guided radiation therapy of pancreatic cancer: 50 successful cases without fluoroscopy. Gastrointest Endosc. 2010 Mar;71(3):513-8. doi: 10.1016/j.gie.2009.10.030. PMID 20189509
- [Background] Farrell JJ, Sherrod A, Parekh D. EUS-guided fine-needle tattooing for preoperative localization of early pancreatic adenocarcinoma. Gastrointest Endosc. 2009 Jan;69(1):176-7. doi: 10.1016/j.gie.2008.03.1069. Epub 2008 Jul 2. No abstract available. PMID 18599051
- [Background] Lennon AM, Newman N, Makary MA, Edil BH, Shin EJ, Khashab MA, Hruban RH, Wolfgang CL, Schulick RD, Giday S, Canto MI. EUS-guided tattooing before laparoscopic distal pancreatic resection (with video). Gastrointest Endosc. 2010 Nov;72(5):1089-94. doi: 10.1016/j.gie.2010.07.023. PMID 21034909